CLINICAL TRIAL: NCT04668768
Title: HM-178: Assessing Methods for Improvement in Methotrexate Toxicity Management and Detection of Central Nervous System Involvement of Aggressive Lymphoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: To be terminated due to slow accrual, patient still in follow up
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-178; 20-1071 (Other: Fox Chase cancer Center)
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — glucarpidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Glucarpidase (Experimental): Prophylactic glucarpidase treatment
  Interventions: Drug: Glucarpidase

INTERVENTIONS:
Drug: Glucarpidase — Glucarpidase injection to prevent toxicities due to high dose methotrexate treatment

SUMMARY:
This is a study to use glucarpidase prophylactically to treat methotrexate induced toxicities in lymphoma patients with cerebral involvement.

DETAILED DESCRIPTION:
Treatment and prophylaxis against CNS (central nervous system) lymphoma typically consist of a regimen containing high dose methotrexate (HD MTX), which requires inpatient monitoring in order to ensure adequate clearance of methotrexate levels (MTX). The goal of this prospective, multi-institution study is to evaluate the effect of prophylactic glucarpidase in patients receiving high dose MTX and are at increased risk of delayed MTX clearance and nephrotoxicity. Glucarpidase is a recombinant bacterial enzyme (carboxypeptidase G2) that can convert MTX to non-cytotoxic metabolites (DAMPA). This is the first controlled trial comparing glucarpidase with supportive care alone in patients with MTX induced nephrotoxicity and delayed MTX clearance.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of Non-Hodgkin Lymphoma and either:

  1. High risk of CNS relapse warranting MTX prophylaxis
  2. Evidence of CNS involvement (either PCNSL or secondary CNS lymphoma) warranting therapeutic MTX treatment
  3. DLBCL

  i. Transformation to DLBCL from an antecedent low-grade lymphoma is permitted d. Burkitt lymphoma (BL) e. Plasmablastic lymphoma f. Blastoid variant of Mantle Cell lymphoma g. Richter Transformation h. Primary CNS Lymphoma i. Secondary CNS lymphoma of any B cell lineage j. B cell Non-Hodgkin Lymphoma with neurologic symptoms suspicious for CNS involvement
* Patients must have at least one of the following 2 criteria;

  1. aged > 65 year with baseline CrCl (creatinine clearance) > 30 ml/min/1.73 m2
  2. any age with a baseline CrCl of 30-59 ml/min/1.73 m2
* Patients must meet criteria for and are appropriate candidates for treatment or prophylaxis with high dose systemic MTX of 3.5 g/m2 if CrCl > 60 ml/min and 2 g/m2 if Cr 30-59 mL/min.
* Patients planned to have 2 or more cycles of high dose MTX as part of treatment regimen. If patents are planned to have more than 4 cycles of MTX, they can be included in study, however glucarpidase will be provided only for up to 4 cycles of MTX.
* Patients must be willing and eligible to undergo diagnostic lumbar puncture for initial staging and also post treatment if evidence of CNS involvement
* Patients with confirmed CNS involvement of disease on lumbar puncture testing or those with clinical symptoms of CNS involvement will require baseline and post treatment brain and spinal MRI. If there is contraindication to MRI, CT scan is permitted.
* Patients must be willing and able to comply with scheduled visits and testing
* Patients must have adequate bone marrow and organ function

  1. Absolute neutrophil count (ANC) >/= 1.0 x 10^9/L
  2. Platelets >/= 100 x 10^9/L and no platelet transfusion within the past 28 days prior to study registration
  3. Hemoglobin (Hgb) >/= 8g/dL and no red blood cells (RBC) transfusion within the past 28 days prior to study registration
  4. International Normalized Ratio (INR) </= 1.5 and PTT (aPTT) </= 1.5 times the upper limit of normal
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 3 times the upper limit of normal
  6. Serum bilirubin </= 1.5 times the upper limit of normal; or total bilirubin </= 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome
  7. CrCl >/= 30 mL/min using the Cockcroft-Gault equation; Men: CrCl (min/mL) = (140-age) X (actual weight in kg) / 72 X serum creatinine (mg/dL); Women: CrCl (mL/min) = (140-age) X (actual weight in kg) X 0.85 / 72 X serum creatinine (mg/dL)
* Patients with therapeutically intervenable ascites fluid and/or pleural effusions are permitted on trial. However, patients must demonstrate absent or mild/trace effusion on post procedure imaging with ultrasound or CT scan within 7 days of each MTX cycle
* Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose.
* Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry

Exclusion Criteria:

* Patients who received CNS directed therapy (intrathecal chemotherapy or systemic HD-MTX) or glucarpidase prior to enrollment. Patients may receive intrathecal prophylaxis at time of initial CSF (cerebrospinal) fluid collection or as part of treatment protocol
* Patients with moderate or severe pleural effusion and/or abdominal ascites at time of enrollment that are not amenable to therapeutic thoracentesis or paracentesis, respectively
* Patients with contraindication or refusal to have cerebrospinal fluid sampling
* Patients with contraindication or refusal to have inpatient HD-MTX administration as part of therapy Patients may not be receiving any other investigational agent
* Patients who will require any medications or substances that are inhibitors or inducers of glucarpidase or MTX during hospitalization for therapy administration are ineligible.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Rate of methotrexate clearance | 6 months
  Number days for methotrexate clearance

SECONDARY OUTCOMES:
Progression free survival | 6 months
  Duration that patients is free of cancer from the time of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States